CLINICAL TRIAL: NCT06827262
Title: Intracept Minimally-invasive PROcedure for VErtebrogenic Back Pain
Acronym: IMPROVE
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: REL025
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Chronic Low-back Pain; Vertebrogenic Pain Syndrome
Keywords: Intraosseous basivertebral nerve ablation; Axial low back pain; Low Back Pain
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Intracept™ Intraosseous Nerve Ablation Systems: Subjects with pain treated with a commercially approved Intracept™ Intraosseous Nerve Ablation System
  Interventions: Device: Intracept™ Intraosseous Nerve Ablation

INTERVENTIONS:
Device: Intracept™ Intraosseous Nerve Ablation — Intracept™ Intraosseous Nerve Ablation for treatment of patients diagnosed with vertebrogenic pain

SUMMARY:
Compile real-world outcomes of commercially approved Intracept™ Intraosseous Nerve Ablation Systems in the treatment of patients diagnosed with vertebrogenic pain.

DETAILED DESCRIPTION:
The objective of this study is to compile real-world outcomes of commercially approved Intracept™ Intraosseous Nerve Ablation Systems in the treatment of patients diagnosed with vertebrogenic pain.

ELIGIBILITY:
Inclusion Criteria:

* Study candidate is scheduled to be treated with a commercially approved Intracept™ Intraosseous Nerve Ablation System per local Instructions for Use (IFU).
* Signed a valid, IRB/EC-approved informed consent form.

Exclusion Criteria:

* Meets any contraindications per locally applicable Instructions for Use (IFU).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are established patients in a medical practice who will receive intraosseous nerve ablation to treat vertebrogenic pain utilizing a commercially approved Intracept™ Intraosseous Nerve Ablation System per local Instructions for Use according to standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2034-07 (Estimated); Study Completion 2034-07 (Estimated)

PRIMARY OUTCOMES:
Change in Disability (Oswestry Disability Index (ODI) from Baseline | 60-months post-procedure
  The Oswestry Disability Index (ODI) is a validated questionnaire of pain-related disability with total score on a scale of 0 (no disability) to 100 (complete disability). Categories for ODI total score are 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The published minimally clinically important difference for change in ODI is 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, M.A., Study Director — Boston Scientific Corporation
Locations (14):
- United States (14):
  - Flagstaff Bone & Joint, Flagstaff, Arizona
  - MarinHealth Spine Institute, Larkspur, California
  - The Spine Wellness Center in Westport, Westport, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - North Idaho Day Surgery, LLC, Post Falls, Idaho
  - Illinois Bone and Joint Institute, Barrington, Illinois
  - Commonwealth Pain and Spine, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - iSpine Clinics, Maple Grove, Minnesota
  - New York Spine and Pain Specialists, Port Jefferson Station, New York
  - University of Rochester, Rochester, New York
  - Pacific Sports and Spine, Eugene, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Utah Orthopaedic Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No